CLINICAL TRIAL: NCT06176352
Title: A Phase III, Multicenter, Randomized, Double-Masked, Active Comparator-Controlled Study to Evaluate the Efficacy and Safety of Faricimab in Patients With Choroidal Neovascularization Secondary to Pathologic Myopia
Brief Title: A Study to Evaluate the Efficacy and Safety of Faricimab in Patients With Choroidal Neovascularization Secondary to Pathologic Myopia
Acronym: POYANG
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR44829; 2023-506707-25-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-12-11; First posted 2023-12-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Choroidal Neovascularization Secondary to Pathologic Myopia
MeSH Terms: interventions — faricimab; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Faricimab (Experimental): All participants randomly assigned to Arm A will receive faricimab 6 mg at Day 1. Once every 4 weeks (Q4W) after Day 1, participants will receive treatment with faricimab on a pro re nata (PRN) basis dependent on prespecified retreatment criteria.
  Interventions: Drug: Faricimab; Procedure: Sham Procedure
- Arm B: Ranibizumab (Active Comparator): All participants randomly assigned to Arm B will receive ranibizumab 0.5 mg at Day 1. Once every 4 weeks (Q4W) after Day 1, participants will receive treatment with ranibizumab on a pro re nata (PRN) basis dependent on prespecified retreatment criteria.
  Interventions: Drug: Ranibizumab; Procedure: Sham Procedure

INTERVENTIONS:
Drug: Faricimab — Faricimab 6 mg intravitreal (IVT) injection on Day 1 with Q4W PRN treatment thereafter to Week 44. At Week 48, participants will attend a follow-up visit.
  Other Names: VABYSMO®; faricimab-svoa; RO6867461; RG7716
  Arms: Arm A: Faricimab
Drug: Ranibizumab — Ranibizumab 0.5 mg intravitreal (IVT) injection on Day 1 with Q4W PRN treatment thereafter to Week 44. At Week 48, participants will attend a follow-up visit.
  Other Names: Lucentis
  Arms: Arm B: Ranibizumab
Procedure: Sham Procedure — The sham is a procedure that mimics an intravitreal (IVT) injection, but involves the blunt end of an empty syringe (without a needle) being pressed against the anesthetized eye. Participants will undergo the sham procedure at study visits where no study drug is to be administered, in order to maintain masking.

SUMMARY:
This is a Phase III, multicenter, randomized, double-masked, active comparator-controlled study evaluating the efficacy and safety of faricimab in patients with myopic choroidal neovascularization (CNV). This non-inferiority study will compare 6.0 mg faricimab versus 0.5 mg ranibizumab administered at a pro-re-nata (PRN) dosing regimen after an initial active IVT treatment administration at randomization (Day 1).

ELIGIBILITY:
Inclusion Criteria:

1. Treatment-naïve choroidal neovascularization (CNV) secondary to myopia
2. Diagnosis of active myopic CNV in the study eye:

   1. Presence of high myopia, worse than -6 diopters of spherical equivalence
   2. Antero-posterior elongation measurement greater than or equal to 26.0 mm
   3. Presence of posterior changes compatible with pathologic myopia (e.g., tessellated fundus, lacquer cracks, etc.)
   4. Presence of active leakage from CNV on FFA (determined by Central Reading Centre [CRC])
   5. Presence of intraretinal or subretinal fluid or increase of CST on OCT (determined by CRC)
3. BCVA of 78 to 24 letters, inclusive (20/32 to 20/320 approximate Snellen equivalent), using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol on Day 1
4. Overtly healthy as determined by medical evaluation that includes medical history, physical examination, and laboratory tests
5. Ability to comply with the study protocol, in the Investigator's judgment
6. Other protocol-defined inclusion criteria apply

Exclusion Criteria:

1. Any major illness or major surgical procedure within 1 month before screening
2. Pregnancy or breastfeeding, or intention to become pregnant during the study or within 3 months after the final study treatment administration
3. Uncontrolled blood pressure (systolic >180 millimetres of mercury [mmHg], diastolic >100 mmHg)
4. Stroke (cerebral vascular accident) or myocardial infarction within 6 months prior to Day 1
5. History of systemic or ocular disease that would contraindicate treatment with the investigational drug or comparator
6. Uncontrolled glaucoma in study eye
7. Any prior or concomitant treatment for CNV or vitreomacular-interface abnormalities, including, but not restricted to, intravitreal, periocular or laser interventions in study eye
8. Prior or concomitant periocular or intravitreal pharmacological treatment, including anti-VEGF medication, for other retinal diseases (e.g. geography atrophy, nAMD, DME etc.) in study eye
9. Other protocol-defined exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Best-Corrected Visual Acuity (BCVA) Averaged Over Weeks 4, 8, and 12 | Baseline and Average of Weeks 4, 8, and 12

SECONDARY OUTCOMES:
Change from Baseline in BCVA Over Time | From Baseline through Week 48
Percentage of Participants Gaining ≥15 Letters in BCVA from Baseline Averaged Over Weeks 4, 8, and 12 | Baseline and Average of Weeks 4, 8, and 12
Percentage of Participants Gaining ≥15 Letters in BCVA from Baseline Over Time | From Baseline through Week 48
Percentage of Participants Avoiding a Loss of ≥15 Letters in BCVA from Baseline Over Time | From Baseline through Week 48
Percentage of Participants Gaining ≥15 Letters in BCVA from Baseline or Achieving a BCVA of ≥84 Letters Over Time | From Baseline through Week 48
Percentage of Participants with BCVA Snellen Equivalent of 20/40 or Better Over Time | From Baseline through Week 48
Percentage of Participants with BCVA Snellen Equivalent of 20/200 or Worse Over Time | From Baseline through Week 48
Percentage of Participants Only Receiving One Injection From Baseline to Weeks 12, 24, and 48 | From Baseline to Weeks 12, 24, and 48
Number of Intravitreal Injections Received From Baseline to Weeks 12, 24, and 48 | From Baseline to Weeks 12, 24, and 48
Change from Baseline in Central Subfield Thickness (CST) of the Study Eye Averaged Over Weeks 4, 8, and 12 | Baseline and Average of Weeks 4, 8, and 12
Change from Baseline in CST of the Study Eye Over Time | From Baseline through Week 48
Change from Baseline in Total Area of the Choroidal Neovascularization Lesion at Weeks 12 and 48 | Baseline, Weeks 12 and 48
Change from Baseline in Total Area of the Choroidal Neovascularization Leakage at Weeks 12 and 48 | Baseline, Weeks 12 and 48
Percentage of Participants with Absence of Macular Leakage at Weeks 12 and 48 | Weeks 12 and 48
Incidence and Severity of Ocular Adverse Events | From first dose until 35 days after the last dose of study treatment (up to 48 weeks)
Incidence and Severity of Non-Ocular Adverse Events | From first dose until 35 days after the last dose of study treatment (up to 48 weeks)
Prevalence of Anti-Drug Antibodies (ADAs) at Baseline and Incidence of ADAs During the Study | At Baseline and from first dose until end of study (up to 48 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (63):
- Australia (4):
  - Strathfield Retina Clinic, Strathfield, New South Wales
  - Sydney Eye Hospital, Sydney, New South Wales
  - Sydney Retina Clinic and Day Surgery, Sydney, New South Wales
  - Centre For Eye Research Australia, East Melbourne, Victoria
- China (17):
  - Beijing Hospital of Ministry of Health, Beijing
  - Beijing Tong Ren Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - The Second Hospital of Jilin University, Changchun
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin
  - Qingdao Eye Hospital of Shandong First Medical University, Qingdao
  - Eye & ENT Hospital of Fudan University, Shanghai
  - Shanghai First People's Hospital, Shanghai
  - First Hospital of China Medical University, Shenyang
  - Shanxi Eye Hospital, Taiyuan
  - Tianjin Medical University Eye Hospital, Tianjin
  - Eye Hospital, Wenzhou Medical University, Wenzhou
  - Central Theater General Hospital of the Chinese People's Liberation Army, Wuhan
  - Wuxi No.2 People's Hospital, Wuxi
  - Xi'an People's Hospital (Xi'an Fourth Hospital), Xi'an
- France (7):
  - Chi De Creteil, Créteil
  - Hopital de la croix rousse, Lyon
  - Centre Paradis Monticelli, Marseille
  - CHU Nantes - Hotel Dieu, Nantes
  - Hopital Lariboisiere, Paris
  - Fondation Rothschild, Paris
  - Centres Ophtalmologique St Exupéry, Saint-Cyr-sur-Loire
- Germany (3):
  - Universitatsklinikum Koln, Cologne
  - Universitätsklinikum Freiburg, Klinik für Augenheilkunde, Freiburg im Breisgau
  - Knappschaftsklinikum Saar GmbH, Sulzbach
- Hong Kong (2):
  - The University of Hong Kong, Hong Kong
  - Hong Kong Eye Hospital, Mong Kok
- Italy (6):
  - Ospedale Clinicizzato SS Annunziata, Chieti, Abruzzo
  - Policlinico di Bari, Bari, Apulia
  - Ospedale Monaldi - AORN dei Colli, Napoli, Campania
  - Fondazione G.B. Bietti Per Lo Studio E La Ricerca in Oftalmologia-Presidio Ospedaliero Britannico, Rome, Lazio
  - Fondazione Irccs Ca' Granda Ospedale Maggiore Policlinico-Clinica Regina Elena, Milan, Lombardy
  - A.O. Universitaria S. Maria Della Misericordia Di Udine, Udine, Veneto
- Poland (6):
  - Klinika Okulistyczna ?Jasne Blonia? Sp. z o. o., ?ód?
  - OFTALMIKA Sp. z o.o, Bydgoszcz
  - Gabinet Okulistyczny Prof Edward Wylegala, Katowice
  - Centrum Medyczne UNO-MED, Krakow
  - Gabinet Okulistyczny Jerzy Mackiewicz, Lublin
  - Centrum Diagnostyki i Mikrochirurgii Oka LENS, Olsztyn
- Singapore (4):
  - National University Hospital, Singapore
  - Singapore Eye Research Institute, Singapore
  - Asia Pacific Eye Centre, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (5):
  - Yeungnam University Medical Center, Daegu
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Kim's Eye Hospital, Seoul
- Spain (6):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Complejo Hospitalario Universitario de Santiago., Santiago de Compostela, LA Coruna
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital de la Arruzafa. Servicio de Oftalmologia, Córdoba
  - Oftalvist, Madrid
- Taiwan (3):
  - Far Eastern Memorial Hospital, New Taipei City
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital, Zhongzheng Dist.

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing